CLINICAL TRIAL: NCT07139184
Title: Risk Factor Analysis for Charcot Foot in Patients With Diabetes Mellitus: The Interplay of Inflammatory Cytokines and Metabolic Factors
Acronym: RFA-CF-DM-ICMF
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Ali Mohamed, Principal Investigator, Assiut University
Other Study IDs: AMAAmrMohammedAli
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Charcot Foot
Keywords: Charcot Foot Diabetes Mellitus TNF alpha IL 10
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The case group: (30 cases): is comprised of patients with diabetes mellitus suffering from Charcot foot and diagnosed clinically.
  Interventions: Diagnostic Test: Diagnosis of Charcot foot disease; Diagnostic Test: Hematologic and biochemical parameters,; Diagnostic Test: ELIZA Assay
- The control group: (30 cases): is comprised DM patients without Charcot foot.
  Interventions: Diagnostic Test: Hematologic and biochemical parameters,; Diagnostic Test: ELIZA Assay

INTERVENTIONS:
Diagnostic Test: Diagnosis of Charcot foot disease — Diagnosis of Charcot foot disease will be obtained from the results of physical examination and according to x-ray examination of foot which was performed at the Radiology Department of Assiut University Hospital. The Eichenholtz classification system, developed by Sidney N. Eichenholtz in 1966, categorizes Charcot arthropathy (also known as Charcot foot) into three stages based on clinical and radiographic findings. These stages are development, coalescence, and reconstruction
  Groups: The case group: (30 cases)
Diagnostic Test: Hematologic and biochemical parameters, — Hematologic and biochemical parameters, including lymphocyte, monocyte, neutrophil, and platelet counts, as well as glucose, HbA1c, triglyceride (TG), HDL, and LDL levels, will be extracted from patient records.
  NLR=absolute neutrophil count (109/L)/absolute lymphocyte count (109/L), PLR=platelet count (109/L)/absolute lymphocyte count (109/L), LMR=absolute lymphocyte count (109/L)/absolute monocyte count (109/L), GLR=glucose (mg/dL)/absolute lymphocyte ratio (109/L), TGR=triglyceride (mg/dL)/glucose ratio (mg/dL), THR=triglyceride (mg/dL)/HDL ratio (mg/dL), SIRI = absolute neutrophil count (109/L) × absolute monocyte count (109/L)/ absolute lymphocyte count (109/L), SII = platelet count (109/L) × absolute monocyte count (109/L)/absolute lymphocyte count (109/L), TyG index = fasting triglyceride (mg/dL) × fasting plasma glucose (mg/dL)/2, PIV =absolute neutrophil count (109/L) × platelet count (109/L) × absolute monocyte count (109/L)/absolute lymphocyte count (109/L).
Diagnostic Test: ELIZA Assay — For each patient, 2 ml of blood will be obtained. The serum levels of IL-10, TNF-α will be assessed by using (ELISA) kit obtained from (Biodiagnostic company, Egypt) according to the manufacturer protocol.

SUMMARY:
Diabetes mellitus (DM) is among the most common metabolic disorders globally. According to the data from international research, the number of persons with diabetes mellitus reached 366 million in 2011 and is predicted to increase to 552 million by 2030.

DETAILED DESCRIPTION:
Hyperglycaemia is a hallmark of diabetes mellitus resulting from defects in insulin secretion, insulin action, or both. Diabetes-related chronic hyperglycaemia is linked to long-term harm complications and failure of several organs, particularly the heart, blood vessels, kidneys, eyes, and nerves and even the musculoskeletal system Charcot neuroarthropathy, is a condition that develops in people with diabetes and neuropathy, causing damage to the bones and joints in the foot There are several risk factors for developing Charcot foot in patients with DM, such as age, gender, duration of diabetes mellitus, blood pressure, blood lipid levels, smoking, and levels of HbA1c. However, little is known about the most significant risk factor to develop such debilitating Charcot foot disease.

Acute Charcot arthritis is also characterized by a marked inflammatory response. Several chronic pro-inflammatory markers are elevated in affected individuals including interleukin-1β, interleukin 6, and tumour necrosis factor-α, and increased receptor activation of nuclear factor-K β ligand, which is imbalanced with its receptor and osteoprotegerin.

Interleukin-10 (IL-10) is a multifunctional cytokine that plays a key role in controlling inflammation and preserving cellular balance. Its primary function is anti-inflammatory, helping to prevent excessive immune reactions by acting mainly through the Jak1/Tyk2 and STAT3 signaling pathway. However, IL-10 can also act as an immune activator under certain conditions, showing stimulatory effects that support immune responses in specific conditions. Given the pivotal role of IL-10 in immune modulation, this cytokine could have relevant implications in pathologies characterized by hyperinflammatory state such as Charcot foot disease.

TNF-α is a member of the vast cytokine family being considered a proinflammatory substance produced many by macrophages and other cells belonging to the innate immunity, many of them classified as indeed Antigen Presenting Cells (APCs) involved in the complex chemotactic process of activation of the adaptive immunity. Elevated levels of TNF-α have been implicated in the development and progression of various neuropathies, including those associated with diabetes.

Although Charcot foot disease is a frequent complication of diabetic neuropathy, less is known about the possibility of its early prevention. This research aims to highlight potentially important early identifiable biomarkers that can lead to Charcot foot disease in patients with DM.

ELIGIBILITY:
Inclusion . Inclusion criteria:

* Adult Patients who are diagnosed with DM who are willing to participate in the study with informed consent form.

  b. Exclusion criteria:
* Patients with neuritis / neuropathy of the lower extremity due to other causes other than DM
* Significant trauma that may cause peripheral nerve damage.
* Patient with routine use of corticosteroid
* Previous history of smoking
* Patients with chronic renal impairment due to diseases other than DM (creatinine > 1.4 mg/dL), previous myocardial infarction or stroke, history of cancer.
* Patients with iron deficiency anemia or uremia affecting HbA1c levels or elevated triglyceride or bilirubin levels.
* Patients diagnosed with neurological disease, malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients' data and medical conditions (name, age, gender, occupation, residence, smoking habits, use of corticosteroids, long history of diabetes mellitus, and other diseases such as hyperlipidemia, hypertension, foot and ankle fracture, and peripheral artery disease) were obtained from the Outpatient Clinic in Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The study will investigate the role of IL-10 and TNF-alpha as novel biomarkers for early detection of acute Charcot foot disease. | one year
  The study will investigate the role of IL-10 and TNF-alpha as novel biomarkers for early detection of acute Charcot foot disease.

SECONDARY OUTCOMES:
The current work will demonstrate the role of inflammatory markers, glycaemic control, lipid profile, and several other risk factors to predict the occurrence of Charcot foot disease. | one year
  The current work will demonstrate the role of inflammatory markers, glycaemic control, lipid profile, and several other risk factors to predict the occurrence of Charcot foot disease.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roglic G. WHO Global report on diabetes: A summary. International Journal of Noncommunicable Diseases. 2016;1(1):3-8.
- [Background] Silva LB, dos Santos Neto AP, Maia SMAS, dos Santos Guimarães C, Quidute IL, Carvalho AdAT, et al. The Role of TNF-α as a Proinflammatory Cytokine in Pathological Processes. The Open Dentistry Journal. 2019;13:332-8.
- [Background] Pratistha I, Kawiyana K, Aryana W. Duration of Type II DM, HbA1C Levels, TNF-α and IL-10 as Risk Factors for Level Charcot Joint Foot and Ankle in Type II DM Patients. International Journal of Health Sciences and Research. 2022;12:147-56.
- [Background] Uslu MF, Yilmaz M. Are Inflammatory Markers Important for Assessing the Severity of Diabetic Polyneuropathy? Medicina (Kaunas). 2025 Feb 25;61(3):400. doi: 10.3390/medicina61030400. PMID 40142211
- [Background] Rosenbaum AJ, DiPreta JA. Classifications in brief: Eichenholtz classification of Charcot arthropathy. Clin Orthop Relat Res. 2015 Mar;473(3):1168-71. doi: 10.1007/s11999-014-4059-y. Epub 2014 Nov 21. No abstract available. PMID 25413713
- [Background] Garcia-Dominguez M. The Role of TNF-alpha in Neuropathic Pain: An Immunotherapeutic Perspective. Life (Basel). 2025 May 14;15(5):785. doi: 10.3390/life15050785. PMID 40430212
- [Background] Carlini V, Noonan DM, Abdalalem E, Goletti D, Sansone C, Calabrone L, Albini A. The multifaceted nature of IL-10: regulation, role in immunological homeostasis and its relevance to cancer, COVID-19 and post-COVID conditions. Front Immunol. 2023 Jun 8;14:1161067. doi: 10.3389/fimmu.2023.1161067. eCollection 2023. PMID 37359549
- [Background] Bobirca A, Musetescu AE, Bordianu A, Pantea Stoian A, Salmen T, Marinescu DC, Alexandru C, Florescu A, Radu R, Isac S, Patrascu T, Serban D, Bobirca F. Novel Biomarkers Predictive of Diabetic Charcot Foot-An Overview of the Literature. Life (Basel). 2022 Nov 21;12(11):1944. doi: 10.3390/life12111944. PMID 36431079
- [Background] Schmidt BM. Clinical insights into Charcot foot. Best Pract Res Clin Rheumatol. 2020 Jun;34(3):101563. doi: 10.1016/j.berh.2020.101563. Epub 2020 Jul 5. PMID 32641254
- [Background] Dardari D. An overview of Charcot's neuroarthropathy. J Clin Transl Endocrinol. 2020 Oct 28;22:100239. doi: 10.1016/j.jcte.2020.100239. eCollection 2020 Dec. PMID 33251117
- [Background] Casadei G, Filippini M, Brognara L. Glycated Hemoglobin (HbA1c) as a Biomarker for Diabetic Foot Peripheral Neuropathy. Diseases. 2021 Feb 22;9(1):16. doi: 10.3390/diseases9010016. PMID 33671807
- [Background] Wukich DK, Schaper NC, Gooday C, Bal A, Bem R, Chhabra A, Hastings M, Holmes C, Petrova NL, Santini Araujo MG, Senneville E, Raspovic KM. Guidelines on the diagnosis and treatment of active Charcot neuro-osteoarthropathy in persons with diabetes mellitus (IWGDF 2023). Diabetes Metab Res Rev. 2024 Mar;40(3):e3646. doi: 10.1002/dmrr.3646. Epub 2023 May 23. PMID 37218537
- [Background] Farmaki P, Damaskos C, Garmpis N, Garmpi A, Savvanis S, Diamantis E. Complications of the Type 2 Diabetes Mellitus. Curr Cardiol Rev. 2020;16(4):249-251. doi: 10.2174/1573403X1604201229115531. No abstract available. PMID 33407062